CLINICAL TRIAL: NCT03521024
Title: Evaluation of Esthetic and Biomechanical Outcome of Maxillary Anterior Single-Tooth Zirconia Implant Supported PEKK Crowns Versus Lithium Disilicate Crowns on PEKK Abutments: Randomized Controlled Trial
Brief Title: Effect of Zirconia Implant Supported PEKK Crowns Versus Lithium Disilicate Crowns on Esthetics
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Lamiaa Said Zaki AbdelSalam Elfadaly, Dr., Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Lamiaa Said Zaki Abd ElSalam
Record Dates: First submitted 2018-04-26; First posted 2018-05-11 (Actual); Last update posted 2018-05-11 (Actual); Status verified 2018-05

CONDITIONS: Tooth Loss
Keywords: Zirconia implants; PEKK crowns; high performance polymer crowns
MeSH Terms: conditions — Tooth Loss | interventions — poly(phthalazine ether sulfone ketone); lithia disilicate

STUDY DESIGN:
Intervention Model Description: Patient will receive a restoration with superior function, esthetics, and quality.
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- lithium disilicate crowns (Active Comparator): lithium disilicate crowns are well documented in the literatures as successful restoration modality.
  Interventions: Other: poly ether ketone ketone; Other: lithium disilicate
- poly ether ketone ketone crowns (Experimental): pekkton
  Interventions: Other: poly ether ketone ketone; Other: lithium disilicate

INTERVENTIONS:
Other: poly ether ketone ketone — Polyetherketoneketone (PEKK) forms a group of high-performance thermoplastic polymers. PEKK shows excellent biocompatibility and exhibits outstanding properties such as high wear resistance and high compressive (246 MPa), flexural (5.0GPa), and tensile strengths (115 MPa). The material is lightweight, allows shock absorption, and can be veneered with various commercially available dental materials
Other: lithium disilicate — well documented in the literatures as successful restoration modality.

SUMMARY:
aim of study is to evaluate esthetic and biomechanical outcome of maxillary anterior single-tooth zirconia implant supported PEKK crowns compared to lithium disilicate crowns on PEKK abutments .

DETAILED DESCRIPTION:
High performance polymers may be a valid alternative to other conventional materials for abutments and crowns over zirconia implants because of their cushioning effect and elastic modulus (5.1GPa), which absorb occlusal forces and avoid overload of the underlying bone from the direct transmission of biting impacts ; which could optimize and preserve osseointegration with time. Zirconia implants with high performance polymers restorations can be considered a good alternative for replacing natural teeth.

For many years lithium disilicate has been the esthetics standard used in Veneers ,Inlays , onlays, occlusal veneers, partial crowns,minimally invasive crowns and Implant superstructures due to its natural-looking tooth colouring and excellent light-optical properties.

Due to the promising esthetics of high performance polymers as it can be veneered with different veneering materials it would successfully restore esthetics.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years
* No active intraoral or systemic disease
* No pregnancy or lactation
* controlled periodontal conditions
* Adequate bone volume to place an implant
* Occlusal function with a natural tooth

Exclusion Criteria:

1. Current pregnancy.
2. Psychiatric disorders.
3. Smokers
4. Poor motivation.
5. Several occlusal parafunction.
6. Persistent intraoral infections.
7. Severe mucosal disease.
8. Active periodontitis.
9. Poor oral hygiene.
10. Lack of occluding dentition at implant rehabilitation level

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Estimated)
Dates: Start 2018-09-15 (Estimated); Primary Completion 2019-06-15 (Estimated); Study Completion 2019-09-15 (Estimated)

PRIMARY OUTCOMES:
Esthetic outcome | 9 month
  measured by pink and white esthetics score

SECONDARY OUTCOMES:
bone resorption | 9 month
  measured by CBCT and measuring unit Housfield Unit(HU)

CONTACTS AND LOCATIONS:
Overall Officials: Lamiaa Abdelsalam, MSc, Principal Investigator — Cairo University

IPD SHARING:
Plan to Share IPD: Undecided